CLINICAL TRIAL: NCT07170449
Title: Investigation of the Relationship Between Ultrasonographic Parameters and Tactile Sensation in Carpal Tunnel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: Sultan Abdulhamid Han
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Ultrasonography; Tactile Sensation
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Patients with carpal tunnel syndrome
  Interventions: Diagnostic Test: Nerve conduction studies; Diagnostic Test: Median nerve ultrasonography; Diagnostic Test: Sensory testing

INTERVENTIONS:
Diagnostic Test: Nerve conduction studies — Upper extremity nerve conduction studies including median-ulnar sensory and motor responses
Diagnostic Test: Median nerve ultrasonography — Median nerve sonographic cross-sectional area and echogenicity measurements
Diagnostic Test: Sensory testing — tactile sensory tests

SUMMARY:
The aim of this study was to investigate the relationship between different ultrasonographic indices used in patients with carpal tunnel syndrome and the level of tactile sensation.

The primary questions the study aimed to answer are:

• To what extent are the ultrasonographic parameters used in the diagnosis of carpal tunnel syndrome related to the level of sensory complaints in the patient?

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compression neuropathy. The etiology of CTS can be related to work, lifestyle, injury, or genetic predisposition. Exposure to vibrations or repetitive forceful angular movements is among the most common causes of CTS. Certain diseases, such as diabetes, pregnancy, and morbidity, are also thought to be associated with an increased risk of developing CTS. It accounts for 90% of all entrapment neuropathies. Its prevalence in the population is between 1% and 5%, and it is three times more common in women. In CTS, complaints related to motor and sensory deficits are observed in the first three fingers innervated by the median nerve and the radial aspect of the fourth finger. Diagnosis is made by corroborating clinical signs and symptoms with electrophysiological findings. However, recently, ultrasound (US) is frequently preferred for the diagnosis of CTS to evaluate the morphological and mechanical properties of the median nerve. US is considered a highly accurate, effective, and cost-effective diagnostic method for the diagnosis of CTS, with a short evaluation time . Sonographic measurements related to CTS can yield values such as the diameter of the nerve at the entrance and exit of the tunnel. CTS presents with a disturbance in tactile input, such as numbness and loss of sensation in the median nerve dermatom. This sensory loss can cause difficulty in using the patient's hand in activities of daily living. Sonography has recently become widely used in CTS patients. The fact that values measured by sonography can provide information about the clinical status of patients can be considered important data for healthcare professionals. Therefore, our study was designed to examine the relationship between sonographic measurements and tactile sensory levels in patients diagnosed with mild to moderate CTS based on electrodiagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* Electrodiagnostic diagnosis of carpal tunnel syndrome with pain, numbness, burning, and tingling consistent with the median nerve dermatomal area lasting at least 6 weeks.
* Literate
* Agree to participate in the study

Exclusion Criteria:

* Concomitant diabetes, systemic inflammatory disease, active infection, and history of malignancy
* Being <18 and >65 years old
* Being illiterate
* Refusing to participate in the study
* Having a disease with neuropathic pain, such as polyneuropathy, radiculopathy, or MS
* Other concomitant upper extremity entrapment neuropathies (e.g., cubital tunnel syndrome)
* Having undergone surgery for carpal tunnel syndrome
* Rheumatoid arthritis, advanced hand osteoarthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed CTS
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
median nerve ultrasound | 3 Months
  Median nerve maximum cross-sectional area measurement at the level of the carpal tunnel (mm²)
Pointed - blunt discrimination test | 3 Months
  The patient is asked to distinguish between a pointed and a blunt tip by touching the median nerve dermatome.
Moved two point discrimination | 3 months
  The patient's finger is touched, starting from the distal tip and moving proximally, and the patient is asked to distinguish between one and two dots. The distance between the last pair of dots the patient can distinguish is noted in mm.
Fixed Two Point Discrimination Test | 3 months
  The patient's finger is touched starting from the distal tip and working proximally, and the patient is asked to distinguish between one and two dots. The distance between the last pair of dots the patient can distinguish is noted in millimeters.
Semmes Weinstein Test | 3 months
  With the patient's eyes closed, monofilament is applied perpendicularly in a steady manner until the filament bends. Use a smooth motion to touch the skin with the filament, bend the filament for a full second, than lift from the skin. Patient raises hand to indicate that the monofilament touch sensation is perceived.
median nerve ultrasound | 3 months
  Median nerve echogenicity at the level of the carpal tunnel (%)
median nerve ultrasound | 3 months
  Median nerve cross-sectional area measurement at the level of the carpal tunnel inlet (mm²)
median nerve ultrasound | 3 months
  Median nerve cross-sectional area measurement at the level of the carpal tunnel outlet (mm²)
median nerve ultrasound | 3 months
  Median nerve cross-sectional area measurement at the level of the pronator quadratus (mm²)

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | 3 Months
  The scale consists of an 11-question Likert-style symptom severity scale and an 8-question functional status scale. The total score is divided by the number of questions to calculate the score. Higher scores are associated with increased symptom severity and poorer functional status.
S-LANSS | 3 Months
  A score of 12 or more out of 24 on a 7-question scale is considered in favor of neuropathic pain.
SF-12 (Short Form-12) | 3 months
  The SF-12 is a practical test consisting of seven questions that examine the life limits of the patient. The questionnaire includes questions aimed at understanding the physical and psychiatric effects. The results of the survey are calculated using two score calculation tools: physical (PCS-12) and mental (MCS-12). The highest score for the PCS-12 is 56.6, while the highest score for the MCS-12 is 60.7. Higher scores are comparable to a state of resilience and recovery, which can be compared to quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Müyesser Cavlak, PhD, Principal Investigator — Sultan Abdülhamit Han Trainin and Educatioal Hospital; Emre Ata, Assoc Prof, Study Chair — Sultan Abdülhamit Han Trainin and Educatioal Hospital
Locations (1):
- Sultan Abdülhamit Han Trainin and Educational Hospital, Üsküdar, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett MI, Smith BH, Torrance N, Potter J. The S-LANSS score for identifying pain of predominantly neuropathic origin: validation for use in clinical and postal research. J Pain. 2005 Mar;6(3):149-58. doi: 10.1016/j.jpain.2004.11.007. PMID 15772908
- [Background] Sezgin M, Incel NA, Serhan S, Camdeviren H, As I, Erdogan C. Assessment of symptom severity and functional status in patients with carpal tunnel syndrome: reliability and functionality of the Turkish version of the Boston Questionnaire. Disabil Rehabil. 2006 Oct 30;28(20):1281-5. doi: 10.1080/09638280600621469. PMID 17083175
- [Background] Multanen J, Ylinen J, Karjalainen T, Ikonen J, Hakkinen A, Repo JP. Structural validity of the Boston Carpal Tunnel Questionnaire and its short version, the 6-Item CTS symptoms scale: a Rasch analysis one year after surgery. BMC Musculoskelet Disord. 2020 Sep 12;21(1):609. doi: 10.1186/s12891-020-03626-2. PMID 32919457
- [Background] Stevens JC. AAEE minimonograph #26: The electrodiagnosis of carpal tunnel syndrome. Muscle Nerve. 1987 Feb;10(2):99-113. doi: 10.1002/mus.880100202. PMID 3821791
- [Background] Fisse AL, Pitarokoili K, Motte J, Gamber D, Kerasnoudis A, Gold R, Yoon MS. Nerve echogenicity and intranerve CSA variability in high-resolution nerve ultrasound (HRUS) in chronic inflammatory demyelinating polyneuropathy (CIDP). J Neurol. 2019 Feb;266(2):468-475. doi: 10.1007/s00415-018-9158-3. Epub 2018 Dec 15. PMID 30554264
- [Background] Wolny T, Linek P. Reliability of two-point discrimination test in carpal tunnel syndrome patients. Physiother Theory Pract. 2019 Apr;35(4):348-354. doi: 10.1080/09593985.2018.1443358. Epub 2018 Feb 26. PMID 29482409
- [Background] Kim JM, Kim MW, Ko YJ. Correlating ultrasound findings of carpal tunnel syndrome with nerve conduction studies. Muscle Nerve. 2013 Dec;48(6):905-10. doi: 10.1002/mus.23841. Epub 2013 Sep 11. PMID 23512486
- [Background] Aboonq MS. Pathophysiology of carpal tunnel syndrome. Neurosciences (Riyadh). 2015 Jan;20(1):4-9. PMID 25630774
- [Background] Yucel H. Factors affecting symptoms and functionality of patients with carpal tunnel syndrome: a retrospective study. J Phys Ther Sci. 2015 Apr;27(4):1097-101. doi: 10.1589/jpts.27.1097. Epub 2015 Apr 30. PMID 25995565